CLINICAL TRIAL: NCT00334542
Title: A Phase II Study of Simvastatin in Women at High Risk for a New Breast Cancer
Brief Title: Simvastatin in Preventing a New Breast Cancer in Women at High Risk for a New Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: J0485; P50CA088843 (NIH); P30CA006973 (NIH); JHOC-J0485 (Other: SKCCC at Johns Hopkins); SKCCC-J0485 (Other: SKCCC at Johns Hopkins); CDR0000477214 (Registry Identifier: NCI PDQ); NA_00041153 (Other: JHM IRB)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Results first posted 2013-06-25 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; ductal breast carcinoma in situ; breast cancer in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Simvastatin (Experimental): Simvastatin 40 mg for 24-28 weeks
  Interventions: Drug: simvastatin

INTERVENTIONS:
Drug: simvastatin — 24-28 weeks of simvastatin
  Other Names: Zocor

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of simvastatin may keep cancer from coming back in women who are at high risk for a new breast cancer after undergoing surgery for ductal carcinoma in situ or stage I, stage II, or stage III breast cancer.

PURPOSE: This phase II trial is studying how well simvastatin works in preventing a new breast cancer in women at high risk for a new breast cancer after undergoing surgery for ductal carcinoma in situ or stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Describe changes from baseline in a panel of biomarkers (high-sensitivity C-reactive protein [hsCRP], lipid profile, circulating estrogens, and contralateral breast density) in women at high risk of developing new breast cancer who have undergone surgical resection for history of ductal carcinoma in situ or stage I-III invasive breast cancer treated with simvastatin.

Secondary

* Correlate changes in the panel of biomarkers with wild-type versus polymorphic 3-hydroxyl-3-methylglutaryl-Coenzyme A (HMG-CoA) reductase in women treated with simvastatin.

Tertiary

* Evaluate methylation status across a panel of genes that are known to be frequently and specifically hypermethylated in ductal carcinoma in situ (DCIS) and invasive breast cancer (estrogen receptor [ER]-α and ER-β, cyclin D2, RAR-β, Twist, RASSF1A, and HIN-1) and correlate change in cumulative methylation with change in hsCRP, lipid profile, contralateral breast density, estrogen concentrations, and pharmacogenetics.
* Measure changes in the phosphoinositide 3'-kinase (PI3K)/protein kinase B (Akt) signaling pathway (Akt and p-Akt) before and after treatment with simvastatin.

OUTLINE: This is a multicenter study. Patients are stratified according to menopausal status (pre- vs post-menopausal).

Patients receive oral simvastatin once daily for 24-28 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection at baseline and at the end of study treatment for pharmacogenetic and biomarker correlative studies. Patients undergo mammography and measurement of breast density of the contralateral breast at baseline and at the end of study treatment.

Quality of life is assessed at baseline and at the end of study treatment.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of histologically confirmed breast cancer, meeting 1 of the following staging criteria:

  * Ductal carcinoma in situ
  * Stage I-III invasive breast cancer
* At least 3 months since completion of all intended local and systemic therapy, including mastectomy or lumpectomy with or without radiotherapy, adjuvant chemotherapy, and/or endocrine therapy

  * May have declined recommended treatment provided all treatment intended/agreed upon by the patient and treating physician was completed ≥ 3 months ago
* At least 1 healthy intact breast

  * No prior radiotherapy or mastectomy
  * Prior biopsies allowed
* Any hormone-receptor status

PATIENT CHARACTERISTICS:

* Female
* Pre- or post-menopausal
* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No active liver disease
* AST and ALT ≤ 3 times upper limit of normal
* Creatinine clearance ≥ 30 mL/min
* No prior hypersensitivity to any 3-hydroxyl-3-methylglutaryl-Coenzyme A (HMG-CoA) reductase inhibitor or any of its components
* No other concurrent infectious, inflammatory, or autoimmune diseases (at the discretion of principal investigator)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No daily alcohol use > 3 standard drinks per day

  * Standard drink defined as 10 grams of alcohol, which is equivalent to 285 mL of beer, 530 mL of light beer, 100 mL of wine, or 30 mL of liquor
* No selective estrogen receptor modulator or aromatase inhibitor within the past 3 months
* No hormone replacement therapy (HRT) within the past 3 months
* No prior estrogen and/or progesterone HRT ≥ 5 years in duration

  * Vaginal estrogen preparations allowed
* No concurrent HRT
* No other cholesterol-lowering drug, including a statin, within the past 3 months
* No concurrent itraconazole, ketoconazole, nefazodone, cyclosporine, HIV protease inhibitors, clarithromycin, erythromycin, mibefradil, carbamazepine, bosentan, chaparral, amiodarone, or verapamil
* No concurrent daily grapefruit juice consumption > 8 ounces per day
* No other concurrent agents or therapies intended to treat or prevent in situ or invasive breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2009-06 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fackler MJ, McVeigh M, Mehrotra J, Blum MA, Lange J, Lapides A, Garrett E, Argani P, Sukumar S. Quantitative multiplex methylation-specific PCR assay for the detection of promoter hypermethylation in multiple genes in breast cancer. Cancer Res. 2004 Jul 1;64(13):4442-52. doi: 10.1158/0008-5472.CAN-03-3341. PMID 15231653
- [Result] Higgins MJ, Prowell TM, Blackford AL, Byrne C, Khouri NF, Slater SA, Jeter SC, Armstrong DK, Davidson NE, Emens LA, Fetting JH, Powers PP, Wolff AC, Green H, Thibert JN, Rae JM, Folkerd E, Dowsett M, Blumenthal RS, Garber JE, Stearns V. A short-term biomarker modulation study of simvastatin in women at increased risk of a new breast cancer. Breast Cancer Res Treat. 2012 Feb;131(3):915-24. doi: 10.1007/s10549-011-1858-7. Epub 2011 Nov 11. PMID 22076478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were required to have good performance status, intact contralateral breast, and be at least 3 months from planned local and systemic adjuvant treatment.
Period: Overall Study
Arm/Group | Simvastatin
Started | 50
Completed | 45
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — New cancer diagnosis | 1

BASELINE CHARACTERISTICS:
Arm/Group | Simvastatin
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 53 [38 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47
  African American | 1
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in a Panel of Biomarkers (High-sensitivity C-reactive Protein [hsCRP], Lipid Profile, and Circulating Estrogens) From Baseline
Time Frame: Baseline and week 24
Population: Paired baseline and post-simvastatin treatment fasting lipid samples were available for 47 participants, including 45 women who completed the study and from two who discontinued the drug prior to the completion of the 24-28 weeks of drug, and are integrated in the intention-to-treat analyses
Measure: Median (95% Confidence Interval); unit: mg/dl
Arm/Group | Simvastatin
Number analyzed (Participants) | 47
mg/dl
  hsCRP | -0.15 [-1 to 0]
  Total cholesterol | -54 [-58.5 to -39]
  High-density lipoprotein cholesterol (HDL) | -1 [-2 to 3]
  Estrogen (estrone sulfate) | -81.5 [-225.5 to -40.5]

2. Primary Outcome: Change in a Panel of Biomarkers (Contralateral Breast Density) From Baseline
Time Frame: Baseline and week 24
Population: Paired baseline and post-simvastatin treatment mammograms for evaluation of breast density were available for 43 participants.
Measure: Median (95% Confidence Interval); unit: percentage of change
Arm/Group | Simvastatin
Number analyzed (Participants) | 43
percentage of change | -0.78 [-2.0 to 1.2]

3. Secondary Outcome: Prevalence of Breast Gene (Estrogen Receptor [ER]-α and ER-β, Cyclin D2, RAR-β, Twist, RASSF1A, and HIN-1) Hypermethylation
Description: Median change in gene promotor methylation (%M) in the contralateral breast of women with breast cancer after six months of therapy
Time Frame: Change from Baseline to week 24
Population: Methylation values at both time points were only evaluable in 17 participants.
Measure: Median (95% Confidence Interval); unit: percent methylation (%M)
Arm/Group | Simvastatin
Number analyzed (Participants) | 17
percent methylation (%M)
  CyclinD2 (CCND2) | 0.5 [-0.68 to 1.97]
  SCGB3A1 | 0 [-1.9 to 2.43]
  TWIST1 | 0.21 [-1.08 to 0.85]
  RASSF1 | 0 [-1.11 to 1.63]
  RARB | -0.08 [-1.72 to 0.23]
  APC | 0.01 [-0.14 to 0.75]
  CMI | -0.42 [-2.14 to 2.92]

4. Secondary Outcome: Prevalence of Akt and p-Akt Activation by Contralateral Core Breast Biopsies
Time Frame: Baseline and week 24
Population: Enough tissue was not collected to assess this outcome measure.
Arm/Group | Simvastatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 28 weeks
Description: Adverse events data were collected during 24-28 weeks of simvastatin administration
Arm/Group | Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 17/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=50)
Constipation (Gastrointestinal disorders) | 7 (7)
Headache (Nervous system disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5) — Generalized muscle pain/weakness
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) — Generalized muscle pain/weakness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No